CLINICAL TRIAL: NCT00696462
Title: The Effect of Forced Air Warming During Cesarean Section on Postoperative Infectious Morbidity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated for lack of funds to initiate study
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Curtis Baysinger, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 70346
Record Dates: First submitted 2008-06-02; First posted 2008-06-12 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Cesarean Section
Keywords: forced-air warming; Bair Hugger; cesarean section; postoperative infection; surgical site infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Patients in Group A will undergo passive warming with a warmed cotton blanket placed over their upper extremities
- B (Active Comparator): Patients in Group B will have a forced-air warming device applied to the upper body above the waist at the 43 degree Celsius setting.
  Interventions: Device: forced-air warming

INTERVENTIONS:
Device: forced-air warming — forced-air warming device
  Other Names: Bair Hugger device
  Arms: B

SUMMARY:
The purpose of this study will be to assess whether forced air warming decreases the rate of surgical site infections following cesarean section.

DETAILED DESCRIPTION:
Given the physiologic and experimental evidence regarding temperature regulation; it remains convincing that forced air warming is protective against the development of SSI. We will set out to prospectively study the effect of forced air warming on patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) female subjects who will undergo cesarean delivery regardless of indication.
* Subjects who have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Patients scheduled to receive prophylactic antibiotic therapy.

Exclusion Criteria:

* Patients who are undergoing a true emergent cesarean section that does not allow placement of the warming devices.
* Patients undergoing general anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
treatment effects on wound infection | As is current standard of care post procedure

SECONDARY OUTCOMES:
treatment effects on endometritis | as is current standard of care post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Curtis L Baysinger, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com